CLINICAL TRIAL: NCT01346943
Title: The Altura AAA Endograft Safety and Feasibility Study For Exclusion of Abdominal Aortic Aneurysms
Brief Title: The Altura Abdominal Aortic Aneurysm (AAA) Endograft Safety and Feasibility Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Altura Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTURA-FIM-1
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal Aortic Aneurysms, AAA
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AAA Stent Graft System (Experimental): Altura Medical AAA Stent Graft System
  Interventions: Device: Altura Medical Abdominal Aortic Aneurysm Stent-Graft

INTERVENTIONS:
Device: Altura Medical Abdominal Aortic Aneurysm Stent-Graft — Altura Medical AAA Stent Graft System
  Other Names: Altura Medical AAA Stent Graft System

SUMMARY:
The purpose of this study is to evaluate the safety of deploying and implanting the Altura Abdominal Aortic Aneurysm (AAA) Endograft in the treatment of abdominal aortic aneurysms in subjects who are candidates for open surgical aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Subject or subject's legal representative understands and has signed an informed consent.
* Infrarenal aneurysmal neck diameter between 18 and 28mm, inclusive.
* Abdominal aneurysm neck angulation < 45 degrees.
* Infrarenal non-aneurysmal neck >/= 15mm in length.
* Abdominal aneurysm >4.5cm and growth >1.0 cm/yr.
* Limited iliac artery tortuosity.
* Iliac artery fixation length of >/= 15mm.
* Iliac artery diameter between 8 and 19 mm, inclusive.
* Iliac artery diameter accessible by a 14 Fr introducer.
* Subject is a candidate for open surgical repair of abdominal aortic aneurysm.
* Patent iliac or femoral arteries access vessels, size and morphology to allow endovascular access of 14 Fr introducer sheaths and catheters.
* Subject has > one year life expectancy.
* Subject is not placed at additional risk while waiting for additional imaging necessary for vascular treatment.
* Subject is American Society of Anesthesiology (ASA) grade 1 through 3, inclusive.
* Subject is able and willing to comply with 30 day, six (6) month, one (1) year and 2 (two) year follow-up.

Exclusion Criteria:

* Subject has an acutely ruptured or leaking or emergent aneurysm.
* Subject has a dissecting aneurysm.
* Subject has a mycotic or infected aneurysm.
* Subject has current vascular injury due to trauma.
* Subject's aneurysm is thoracic or suprarenal.
* Previous surgical or endovascular aneurysm repair for abdominal aortic aneurysm.
* Subject has thrombus, calcification and/or plaque that may compromise sealing
* Subject has had a myocardial infarction within six (6) months prior to enrollment.
* Subject has current angina or other active cardiac condition such as congestive heart failure, untreated or worsening atrial arrhythmia, ventricular arrhythmia, or valvular disease.
* Subject has undergone other major surgery within the 30 days prior to enrollment.
* Subject is pregnant or nursing.
* Known allergy to nitinol or polyester or contrast material that cannot be pretreated.
* Subject is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta.
* Subject has connective tissue disease (e.g., Marfan's syndrome).
* Subject has a bleeding disorder or anemia defined as hemoglobin < 9.0 mg/dL.
* Subject is hypercoagulable.
* Subject is on dialysis or has compromised renal function as reflected by a serum creatinine >2.2 mg/dL.
* Subject has compromised hepatic function as measured by SGPT (ALT) > three (3) times the upper limit of normal.
* Subject has active systemic infection.
* Subject is participating in another research study involving an investigational agent for the treatment of AAA.
* Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment and the procedures and evaluations pre- and post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The rate of major adverse events. | 30 days
  Adverse events defined as the composite endpoint of death, significant blood loss requiring intervention, respiratory failure, myocardial infarction, renal failure, paralysis, stroke, bowel ischemia and/or device migration causing vascular compromise.

SECONDARY OUTCOMES:
Feasibility of device defined by clinical and technical success | 6 months, 1 year and 2 years
  Evaluate the feasibility of using Altura AAA Endograft. Feasibility is comprised of acute clinical and technical success measured at the time of procedure. Long-term safety will be evaluated at 6 months, 1 year and 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Kramer, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (2):
- Pontificia Universidad Catolica De Chile, Santiago, Chile
- Stradins University Hospital, Riga, Latvia